CLINICAL TRIAL: NCT06131645
Title: The IASLC Grading System as a Predictor for EGFR-TKI Therapy in EGFR-mutant Lung Adenocarcinoma
Brief Title: IASLC Grading System as a Predictor for EGFR-TKI Therapy
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Other Study IDs: GRADS-TKI
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IASLC grading system — A cohort of 2160 patients with invasive nonmucinous EGFR-mutant LADCs were retrospectively collected and classified according to the IASLC grading system. The role of IASLC grading system in EGFR tyrosine kinase inhibitor (TKI) therapy selection either as adjuvant or palliative therapy was investigated.

SUMMARY:
The investigators previously validated the grading system proposed by International Association for the Study of Lung Cancer (IASLC) for invasive nonmucinous lung adenocarcinoma (LADC) for its reproducibility, prognostication function and predictive value of adjuvant chemotherapy (ACT). In this exploratory study, the investigators aimed to investigate the role of IASLC grading system in EGFR tyrosine kinase inhibitor (TKI) therapy selection either as adjuvant or palliative therapy.

ELIGIBILITY:
Inclusion Criteria:

* invasive lung adenocarcinoma patients who underwent complete resection with positive EGFR mutations in exons 18-21.

Exclusion Criteria:

* adenocarcinoma in situ (AIS), minimally invasive adenocarcinoma (MIA), invasive mucinous adenocarcinoma and other variants of adenocarcinoma
* patients with pathologic slides unavailable for re-evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2008 to April 2021, we consecutively collected lung adenocarcinoma patients who underwent complete resection at the Department of Thoracic Surgery, Fudan University Shanghai Cancer Center (FUSCC), Shanghai, China. The 8th TNM staging was used in this study. The study included three main subgroups: (1) patients with p-TNM stage Ib-III LADCs received adjuvant EGFR-TKI or chemotherapy (ADJUVANT subgroup, N=620), (2) patients developed post-operative recurrence and treated with either EGFR-TKI or chemotherapy (RECURRENCE subgroup, N=321), and (3) next-generation sequencing (NGS) was carried out which provided co-occurring mutation information (NGS subgroup, N=1158).
Sampling Method: Non-Probability Sample
Enrollment: 2160 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  DFS was defined as time from initiation of surgery to date of first event (recurrence or death)
Progression-free survival | 5 years
  PFS was defined as time from initiation of systemic palliative treatment to date of disease progression or death for 1L treatment of each patient and the initiation time was re-assigned additionally for each drug applied during the treatment history of the patients regardless of line of therapy (all lines)

SECONDARY OUTCOMES:
Overall survival | 5 years
  was defined as time from surgery to date of death resulting from any cause in ADJUVANT subgroup and from 1L systemic palliative treatment assignment to date of death resulting from any cause in RECURRENCE subgroup.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaoqiang Deng, Shanghai, Please Select, China